CLINICAL TRIAL: NCT06123598
Title: Effects of Mental Practice and Therapeutic Exercise in Mild Smokers: a Randomized Controlled Trial
Brief Title: Effects of Mental Practice and Therapeutic Exercise in Mild Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Francisco Martínez Arnau, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-FIS-2731776-2
Record Dates: First submitted 2023-10-06; First posted 2023-11-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Smokers
Keywords: smokers; therapeutic exercise; mental practice; respiratory function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be assigned to one of two study groups by the person conducting the intervention.
  All participants receive mental practice (real or sham) and the exercise program.
  The evaluators are unaware of the assignment at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Action observation plus exercise (Experimental): Therapeutic exercise plus action observation training
  Interventions: Behavioral: Therapeutic exercise program plus action observation training
- Sham observation plus exercise (Sham Comparator): Therapeutic exercise plus sham action observation training
  Interventions: Behavioral: Therapeutic exercise program plus sham action observation training

INTERVENTIONS:
Behavioral: Therapeutic exercise program plus action observation training — Participants make an observation of actions related to the training they are going to perform before each session. Subsequently, they perform the therapeutic exercise program of 6 sessions in a period of 2 weeks.
  Arms: Action observation plus exercise
Behavioral: Therapeutic exercise program plus sham action observation training — Participants make a sham observation before each session. Subsequently, they perform the therapeutic exercise program of 6 sessions in a period of 2 weeks.
  Arms: Sham observation plus exercise

SUMMARY:
The goal of this clinical trial is to learn about the effects who would add mental practice based on action observation to a therapeutic exercise program in young mild smokers.

The main question it aims to answer is whether the observation of actions prior to the implementation of a therapeutic exercise program improves the response to it on respiratory, strength and muscle function variables.

Participants will be assigned to one of 2 study groups:

G1) Therapeutic exercise plus action observation training (n=20) G2) Therapeutic exercise plus sham action observation training (n=20)

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Had a pack per year index of <5 (mild smoking index).

Exclusion Criteria:

Those who presented:

* a respiratory pathology,
* cardiac, systematic, or metabolic disease,
* history of recent surgery,
* vertebral fracture,
* or osteoarticular disorders of the spine area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Respiratory strength | Before the start of the program, in the middle of the program (1 week) and at the end of the program (2 weeks)
  Maximal respiratory pressures (in H2O centimeters)

SECONDARY OUTCOMES:
Spirometric parameters | Before the start of the program, in the middle of the program (1 week) and at the end of the program (2 weeks)
  Forced expiratory volume in the first second FEV1 (in liters/second) and forced expiratory volume FVC (In liters/second) obtained from a spirometry
Physical function | Before the start of the program, in the middle of the program (1 week) and at the end of the program (2 weeks)
  5 times sit-to-stand test (in seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No